CLINICAL TRIAL: NCT00430066
Title: Glivec (Imatinib Mesylate) in the Treatment of Polycythemia Vera
Brief Title: Effects of Imatinib Mesylate in Polycythemia Vera
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571POLIVERA
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib Mesylate (Experimental): 400 mg/day by mouth for 6 months (+ 6 months in case of responsiveness)
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — 400 mg/die for 6 months

SUMMARY:
The purpose of this study is to determine the activity of Glivec 400 mg po daily, as single agent, in inducing a haematological response in Polycythemia Vera.

The patients will be asked to have additional bone marrow and blood samples collected: these samples will be used to evaluate how the disease is responding to the drug.

DETAILED DESCRIPTION:
Hematocrit <45% in men or <42% in women at 1°evaluation within 6 months In case of complete or partial responsiveness, experimental treatment will be continued until 12 months In case of disease progression or treatment failure, experimental drug will be withdrawn and patient will be out of the study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Polycythemia Vera requiring treatment with either phlebotomy or Hydroxyurea
* Age >18 years
* Signed written informed consent form

Exclusion Criteria:

* Pregnancy or breast-feeding
* Creatinine >3 max NV
* Bilirubin >3 max NV
* AST/ALT >3 max NV
* Concomitant and severe psychiatric disorder
* Concomitant neoplastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Reduction of Haematocrit to less than 45%. | 6-12 months

SECONDARY OUTCOMES:
Response duration | 6-12 months
Safety profile | 6-12 months
Reduction in platelet count and spleen size | 6-12 months
Reduction of incidence phlebotomies. | 6-12 months
Symptoms improvement in patients. | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Enrica Morra, MD, Study Director — Divisione di Ematologia - Ospedale Niguarda Ca' Granda